CLINICAL TRIAL: NCT01029145
Title: Non-interventional Study to obSERve currENt Management of Index Episode in Patients With Bipolar Disorder Treated bY Seroquel XR
Brief Title: Management of Index Episode in Patients With Bipolar Disorder Treated by Seroquel XR
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca PHARMA SRL ROMANIA
Other Study IDs: NIS-NRO-SER-2009/1
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2010-09-20 (Estimated); Status verified 2010-09

CONDITIONS: Bipolar Disorder; New Occurred Episode
Keywords: Bipolar disorder; New occured episode: manic depressive or mixed
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Bipolar patients that experience a new episode of any type

SUMMARY:
The primary purpose of the study is to explore management of symptomatology in patients with bipolar disorder that experience a new manic,depressive or mixed episode and are treated with Seroquel XR monotherapy/adjuctive, in routine clinical practice in Romania

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for entry into the study, male and females, will have a diagnosis of bipolar disorder, as defined by DSM-IV-TR and the current episode, whether it is manic, depressed or mixed will be treated with Seroquel XR since 1 week before entering the programme.
* All eligible patients will be included in the programme provided they will receive information in advance and will sign consent to grant access to the data collected with regard to their condition during the observation interval proposed.

Exclusion Criteria:

* All the patients who have a known hypersensitivity to Seroquel XR/quetiapine or any of its excipients will not be included in this study.
* Concomitant medication, that could result in drug interactions and could jeopardize patient safety will be carefully considered before having the patient enrolled. Additionally, all precautions applicable for special category patients will be taken into account, as detailed in current valid Romanian SmPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The programme will include patients with bipolar disorder currently experiencing a manic, mixed or depressed episode( named in the protocol the index episode) treated with Seroquel XR for 1 week
Sampling Method: Probability Sample
Enrollment: 537 (Actual)
Dates: Start 2009-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Symptoms severity | 10 weeks ( 4 times:baseline; at 2 weeks; 6 weeks;10 weeks )

SECONDARY OUTCOMES:
QoL/ quality of life | twice in 10 weeks ( v1 and v4)

CONTACTS AND LOCATIONS:
Overall Officials: Ozana Serban, Study Director — AstraZeneca
Locations (30):
- Romania (30):
  - Research Site, Arad, Arad
  - Research Site, Piteşti, Argeş
  - Research Site, Bacau, Bacău
  - Research Site, Bistriţa, Bistrița-Năsăud County
  - Research Site, Botoșani, Botoșani County
  - Research Site, Brăila, Brăila County
  - Research Site, Bucharest, București
  - Research Site, Cluj-Napoca, Cluj Napoca
  - Research Site, Turda, Cluj Napoca
  - Research Site, Palazu Mare, Constanța County
  - Research Site, Craiova, Dolj
  - Research Site, Târgovişte, Dâmbovița County
  - Research Site, Galati, Galați County
  - Research Site, Giurgiu, Giurgiu County
  - Research Site, Tg Jiu, Gorj County
  - Research Site, Miecurea Ciuc, Harghita County
  - Research Site, Hunedoara, Hunedoara County
  - Research Site, Iași, Iaşi
  - Research Site, Luduş, Mureș County
  - Research Site, Oradea, Oradea
  - Research Site, Piatra Neamţ, Piatra Neamt
  - Research Site, Câmpina, Prahova
  - Research Site, Ploieşti, Prahova
  - Research Site, Satu Mare, Satu Mare County
  - Research Site, Suceava, Suceava
  - Research Site, Tg Mures, Tg Mures
  - Research Site, Lugoj, Timisoara
  - Research Site, Timișoara, Timisoara
  - Research Site, Tulcea, Tulcea County
  - Research Site, Rm Valcea, Vâlcea County